CLINICAL TRIAL: NCT01136863
Title: Felodipine Event Reduction Study
Acronym: FEVER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese Academy of Medical Sciences (Other)
Collaborators: Shanxi Kangbao Pharmaceutical company (Unknown); Beijing Hypertension League Insititute (Unknown)
Responsible Party: Lisheng Liu/professor, Fu Wai Hospital, CAMS & PUMC
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 96-906-02-11
Record Dates: First submitted 2010-06-02; First posted 2010-06-04 (Estimated); Last update posted 2010-06-25 (Estimated); Status verified 2005-01

CONDITIONS: Hypertension
Keywords: hypertension; felodipine; moderate to high risk patients
MeSH Terms: conditions — Hypertension | interventions — Felodipine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- felodipine group, active, pill (Active Comparator): felodipine and HCTZ treatment group
  Interventions: Drug: Felodipine
- placebo, no treatment, pill (Placebo Comparator): placebo and HCTZ group
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Felodipine
  Arms: felodipine group, active, pill
Drug: Placebo
  Arms: placebo, no treatment, pill

SUMMARY:
FEVER is an investigator-designed, prospective, multicentre,double-bind, randomized, placebo-controlled,parallel-group trial. The primary objective is to compare the long-term effects on the incidence of fatal and non-fatal stroke (and secondarily of other cardiovascular events) of administering a small dose of the calcium antagonist felodipine (5 mg once a day) or of a placebo, in hypertensive patients whose blood pressure had preliminarily been reduced by administering a low-dose diuretic (hydrochlorothiazide,12.5 mg once a day) to be continued in association with felodipine or placebo, throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

* SBP of 210 mmHg or less and DBP less than 115 mmHg if under antihypertensive treatment; SBP 160-210 mmHg or DBP 95-115 mmHg if untreated. Presence of at least one or two risk factors or cardiovascular diseases Informed consent obtained

Exclusion Criteria:

stroke or myocardial infarction during the previous 6 months; secondary hypertension; unstable angina; cardiomyopathy or significant valvular disease; serum creatinine greater than 178 mmol/l (2.0 mg/dl); gout; uncontrolled diabetes(fasting plasma glucose > 10 mmol/l, 180 mg/dl despite therapy); serious pulmonary or hepatic disease; known contraindications to study drugs; unwillingness to cooperate

Ages: 50 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9800 (Actual)
Dates: Start 1998-04; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
Composite of fatal and non-fatal stroke | During the study period

SECONDARY OUTCOMES:
all cause death | during the study period
cardiac event | during the study period
All cardiovascular events | during the study period
new onset diabetes | during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Lisheng Liu, MD, Principal Investigator — Fu Wai Hospital
Locations (1):
- Fu Wai Hospital, Beijing, China

REFERENCES:
- [Derived] Zhang Y, Zhang X, Liu L, Zanchetti A; FEVER Study Group. Is a systolic blood pressure target <140 mmHg indicated in all hypertensives? Subgroup analyses of findings from the randomized FEVER trial. Eur Heart J. 2011 Jun;32(12):1500-8. doi: 10.1093/eurheartj/ehr039. Epub 2011 Feb 22. PMID 21345850